CLINICAL TRIAL: NCT03266731
Title: Role of Anti-platelet in Treatment of Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Tharwat, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROAITOAIS
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of aspirin and clopidogrel (Experimental)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — evaluates the safety and efficacy of clopidogrel and aspirin as an alternative treatment in patients not eligible for recombinant tissue plasminogen activator or any other acute reperfusion therapy with acute ischemic stroke (AIS) and transient ischemic attack (TIA) within 24 hours of symptoms onset
  Other Names: clopidogrel

SUMMARY:
Role of anti-platelet in treatment of acute ischemic stroke to determine the safety of immediate anti-platelet therapy .that is started as soon as possible within the first 24 hours of the onset of symptoms.

DETAILED DESCRIPTION:
In 2015, stroke was the second most frequent cause of death after coronary artery disease, accounting for 6.3 million deaths (11% of the total).Studies have reported a 30-day recurrence rate of 1.1 to 15 % after stroke and as high as 17% after transient ischemic attack .Therefore, early initiation of antiplatelet agents in ischemic stroke and patients is important to prevent stroke recurrence and is tracked as a quality measure by organizations that accredit stroke centers . Intravenous thrombolysis with alteplase is the mainstay medical treatment for acute ischemic stroke. given intravenously within 4.5 hours of symptom onset, to reopen occluded intracerebral arteries. As in fact most patients with ischemic stroke present to the emergency department beyond the approved time window for thrombolytic or other revascularization therapies beside their high cost and at this time, there are no approved urgent therapies for most of these patients In addition, those who present with rapidly resolving deficit or low National Institutes of Health stroke scale score are generally not considered for thrombolytic treatment, although approximately one third of them may be at high risk for neurological deterioration and recurrent vascular events.This study will evaluates the safety and efficacy of clopidogrel and aspirin in treatment of patients not eligible for recombinant tissue plasminogen activator or any other acute reperfusion therapy with acute ischemic stroke and transient ischemic attack within 24 hours of symptoms onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the patients is 40 years or older.
2. Patients not eligible for recombinant tissue plasminogen activator or any other acute reperfusion therapy presenting after 6hours of onset of symptoms.
3. Patients presented with clinical symptoms of acute stroke or TIA with onset less than 24 hours before starting any treatment.
4. The diagnosis of stroke or TIA basing on clinical examination using National Institute of Health stroke scale (NIHSS) by a stroke specialist

Exclusion Criteria:

1. Any history of ICH or systemic hemorrhage.
2. Any evidence of hemorrhage on baseline CT brain imaging.
3. Patients presented with failed medical or surgical thrombectomy.
4. International normalized ratio (INR) more than 1.5.
5. History of allergy to aspirin or clopidogrel or both of them.
6. Platelets count less than 100,000/mm3.
7. Hematocrit less than 30 mg/dL .
8. glucose less than 50 mg/dL or greater than 400 mg/dL.to exclude hypoglycemia induced focal neurological deficit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-04 (Estimated); Primary Completion 2019-01-04 (Estimated); Study Completion 2020-01-04 (Estimated)

PRIMARY OUTCOMES:
A clinically significant neurologic deterioration | 24 hours
  NIHSS score to detect the outcome of the patients as a greater than or equal to 2-point decrease or a score of 0.

IPD SHARING:
Plan to Share IPD: Undecided